CLINICAL TRIAL: NCT00711165
Title: The Effects of Mometasone on Markers of Airway Inflammation
Brief Title: Mometasone and Markers of Airway Inflammation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Thomas B. Casale, MD, Creighton University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Mometasone TBC
Record Dates: First submitted 2008-07-03; First posted 2008-07-08 (Estimated); Last update posted 2008-07-08 (Estimated); Status verified 2008-07

CONDITIONS: Asthma
Keywords: Asthma; Nitric Oxide; Exhaled Breath Condensate; Methacholine Challenge
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo, 2 puffs, bid
  Interventions: Drug: Placebo
- Memetasone (Experimental): Mometasone
  Interventions: Drug: Mometasone Furoate

INTERVENTIONS:
Drug: Placebo — 2 puffs, qd
  Arms: Placebo
Drug: Mometasone Furoate — 400 mcg, qd for 8 weeks
  Other Names: asmanex
  Arms: Memetasone

SUMMARY:
A post-marketing study to look at the effects of Asmanex on markers of airway inflammation.

DETAILED DESCRIPTION:
Patients with asthma and not treated with anti-inflammatory medications were studied. This was a parallel, randomized, placebo-controlled study to investigate the effects of Asmanex on markers of airway inflammation including exhaled nitric oxide, airway reactivity, FEV1 and nitrates/nitrites and pH in exhaled breath condensate.

ELIGIBILITY:
Inclusion Criteria:

* Asthma
* non-smoker
* FEV1 of at least 60% predicted

Exclusion Criteria:

* Pregnancy or lactation
* Corticosteroid use in past 30 days

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2005-08; Primary Completion 2006-04 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Exhaled Nitric Oxide | 8 weeks

SECONDARY OUTCOMES:
Airway Reactivity | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas B Casale, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Mehta V, Stokes JR, Berro A, Romero FA, Casale TB. Time-dependent effects of inhaled corticosteroids on lung function, bronchial hyperresponsiveness, and airway inflammation in asthma. Ann Allergy Asthma Immunol. 2009 Jul;103(1):31-7. doi: 10.1016/S1081-1206(10)60140-8. PMID 19663124